CLINICAL TRIAL: NCT07167641
Title: Caring for the Carer
Acronym: CFC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Department of Health and Human Services (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-1695
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Care Burden; Care Giving Burden; Caregiver Burnout; Caregiver Wellbeing
Keywords: Cognitive Behavioral Therapy; Supporters; Caregiving; Caregiver Support
MeSH Terms: conditions — Caregiver Burden | interventions — Cognitive Behavioral Therapy; Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caring for the Carer Participants (Experimental): Participants (caregivers and supporters) will participate in four foundational sessions (orientation, goal-setting) and up to 16 CBT-focused sessions. A maximum of 20 individual therapy sessions will be delivered to all participants from their date of enrollment up to 6 months.
  Interventions: Other: Cognitive Behavioral Therapy for Caregivers

INTERVENTIONS:
Other: Cognitive Behavioral Therapy for Caregivers — The intervention includes four "Foundational Sessions" delivered to all participants: Orientation and Engagement, Narrative Exploration, and Goal Setting Sessions at the beginning of treatment, followed by a structured Closing Session at the end of treatment. Beyond the four foundational sessions, caregiver clients complete an additional module based on their top area of need. These modules are called "Core Sessions" and are selected through a collaborative process that draws on caregiver preferences, clinical judgment, and assessment results to ensure treatment is tailored to each caregiver's unique experiences, interests, and goals.

SUMMARY:
The purpose of the present study is to investigate the acceptability and feasibility of implementing a novel, Cognitive Behavioral Therapy (CBT) intervention to caregivers and supporters of individuals who have experienced psychosis, regardless of their relative's engagement in treatment specific to psychosis (i.e., coordinated specialty care (CSC) services). Additionally, the investigators will assess the secondary aim of impact on well-being as a result of the intervention.

DETAILED DESCRIPTION:
Purpose: The purpose of the present study is to investigate the acceptability and feasibility of implementing a novel, Cognitive Behavioral Therapy (CBT) intervention to caregivers and supporters of individuals who have experienced psychosis, regardless of their relative's engagement in treatment specific to psychosis (i.e., coordinated specialty care (CSC) services). Additionally, the investigators will assess the secondary aim of impact on well-being as a result of the intervention.

Participants: 30 caregivers or supporters of individuals who have experienced psychosis and have been referred to or are actively engaged in treatment with two CSC clinics (OASIS and Encompass) Procedures (methods): All participants will be recruited on a rolling basis from two CSC clinics. Participants will engage in a novel, CBT therapy intervention co-developed by Kelsey Ludwig, PhD, and David Penn, PhD. Participants will receive the individual therapy intervention once per week or bi-weekly, for 20 sessions, over the course of 6 months. All therapy sessions will be conducted by trained Masters' or Doctorate level therapists and will be recorded to score treatment fidelity for each therapist. Experiences, wellbeing, and support measures will be taken at baseline and post-treatment, participants will be compensated for these assessments.

ELIGIBILITY:
Inclusion Criteria:

* The participants must be a parent, caregiver, or supporter of a young person who has been referred to a CSC program for First Episode Psychosis (FEP) in the past 3 years. A parent or supporter is considered eligible for the study if their young person was referred to the program but chose not or was unable to engage in CSC or is currently on the waitlist for FEP treatment.
* Parent, caregiver, or supporter must be at least 18 years of age
* Participants recruited from UNC CSC programs
* Parent, caregiver, or supporter must be able to engage in research assessments and consent to audio recording sessions for fidelity ratings

Exclusion Criteria:

* Parent, caregiver, or supporter is currently engaged in legal action against the loved one receiving services/experiencing psychosis
* Parent, caregiver, or supporter's loved one has never experienced psychosis
* Parent, caregiver, or supporter does not speak English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change in the Experience of Caregiving (ECI) Score | Baseline, Month 6
  The Experience of Caregiving (ECI) Scale is a 66-item scale. Answers are on a 5-point scale starting at 0 with options "never," "rarely," "sometimes," "often," and "nearly always". Possible scores range from 0 to 264. Higher scores indicate greater feelings of preparedness for caregiving whereas lower scores reflect feeling less prepared to provide caregiving.
Mean Change in UCLA Loneliness Scale Score | Baseline, Month 6
  The UCLA Loneliness scale is a 20-item scale. Answers are on a 4-point scale with options "I often feel this way," "I sometimes feel this way," "I rarely feel this way," and "I never feel this way." Possible scores range from 20 to 80. Higher scores reflect worse outcomes (greater feelings of loneliness). The UCLA Loneliness Scale is a part of the PhenX Toolkit.
Mean Change in Modified PTSD Checklist for DSM-5 | Baseline, Month 6
  The Modified PTSD Checklist for DSM-5 is a 38-item scale. Answers are on a 5-point scale starting at 0 with options "not at all," "a little bit," "moderately," "quite a bit," and "extremely." Possible scores range from 0 to 80. Higher scores indicate a greater severity of PTSD symptoms.
Mean Change in the Patient Health Questionnaire-8 Score | Baseline, Month 6
  The Patient Health Questionnaire-8 (PHQ-8) is an 8-item scale. Answers are on a 4-point scale ranging from 0 "not at all" to 3 "nearly every day." Possible scores range from 0 to 24. Higher scores reflect worse outcomes (more depressive symptoms).
Mean Change in the General Anxiety Disorder-7 Score | Baseline, Month 6
  The General Anxiety Disorder-7 (GAD-7) is a 7-item scale. Answers are on a 4-point scale ranging from 0 "not at all" to 3 "nearly every day." Possible scores range from 0 to 21. Higher scores reflect worse outcomes (more symptoms of anxiety).
Mean Change in the Self-Compassion Scale Short Form | Baseline, Month 6
  The Self-Compassion Scale Short Form (SCS-SF) is a 12-item scale. Answers are on a 5-point scale ranging from 1 "almost never" to 5 "almost always." Possible scores range from 12-60, with higher scores reflecting higher self-compassion.
Mean Change in Working Alliance Inventory Short Revised | Baseline, Month 6
  The Working Alliance Inventory Short Revised (WAI-SR) is a 12-item scale. Answers are on a 5-point scale ranging from 1 "seldom" to 5 "always." Possible scores range from 12-60, with higher scores indicating greater feelings of alliance between participant and clinician.
Number of Participants Withdrawn or Discontinued | Up to 6 months
  The number of participants who withdraw or discontinue from the study before completing all therapy sessions and providing complete data.
Percentage of Referred Participants Who Enroll | Up to 6 Months
  The percent of potential participants who are referred that enroll, complete all therapy sessions, and provide complete data.

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey A Ludwig, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No